CLINICAL TRIAL: NCT02425319
Title: Motion Analysis of the Proximal Interphalangeal Joint in Healthy Hands, as Well as in Osteoarthritis Hands Following Implantation With the New CapFlex-PIP© Implant Compared With Silicone Implants
Brief Title: CapFlex-PIP© Motion
Status: Completed | Type: Observational
Sponsor: Schulthess Klinik (Other)
Responsible Party: Principal Investigator, Stephan Schindele, Dr. med., Schulthess Klinik
Other Study IDs: CapMotion
Record Dates: First submitted 2015-04-20; First posted 2015-04-23 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Finger Joint; Arthroplasty; Replacement; Motion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- patients with CapFlex-PIP© implant
- patients with silicone implant
- patients with healthy PIP joints

SUMMARY:
The purpose of this study is to describe and to compare the motion analysis parameters, i.e. motion and stability of proximal interphalangeal joints, which were treated with a CapFlex-PIP© implant or silicone implant and to generate basic knowledge about motion analysis of untreated healthy hands.

ELIGIBILITY:
Inclusion Criteria:

* Patients with proximal interphalangeal joint osteoarthritis in the index or middle finger, treated with a CapFlex-PIP© implant or with a silicone implant and with a follow-up time between 12 and 60 months after primary implantation or
* Patient with one untreated healthy hand without joint osteoarthritis
* Patient aged 50 years and over
* Patient willing and able to give written informed consent to participate in the study

Exclusion Criteria:

* Inflammatory disease (e.g. rheumatoid arthritis)
* Pregnant women
* German language barrier to complete the questionnaires
* Any disease process that would preclude accurate evaluation (e.g. neuromuscular, psychiatric or metabolic disorder)
* Legal incompetence
* Participation in any other medical device or medicinal product study within the previous months that could influence the results of the present study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with proximal interphalangeal joint osteoarthritis in the index or middle finger, treated with a CapFlex-PIP© implant or with a silicone implant and with a follow-up time between 12 and 60 months after primary implantation or patient with one untreated healthy hand without joint osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Active PIP joint range of motion (flexion and extension lag) during motion analysis | 1-5 years postoperative
Lateral stability in coronal plane (to ulnar and radial side) during motion analysis | 1-5 years postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Schulthess Klinik, Zurich, Switzerland